CLINICAL TRIAL: NCT00327054
Title: Effectiveness of Nigella Sativa (Kalonji) Seed in Dyslipidemia: A Randomized Controlled Trial
Brief Title: Effectiveness of Nigella Sativa (Kalonji) Seed in Dyslipidemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aga Khan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 05201MED(Grant Fund#1VJ)
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2007-04

CONDITIONS: Hypercholesterolemia; Hypertension; Diabetes Mellitus; Metabolic Syndrome X
Keywords: Dyslipidaemia; Herbal medicine; Home remedy; Alternative medicine; Metabolic syndrome
MeSH Terms: conditions — Hypercholesterolemia; Hypertension; Diabetes Mellitus; Metabolic Syndrome; Dyslipidemias | interventions — Nigella sativa oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nigella sativa seed (Experimental)
  Interventions: Drug: Nigella sativa seed
- Control (No Intervention)

INTERVENTIONS:
Drug: Nigella sativa seed
  Arms: Nigella sativa seed

SUMMARY:
This is a pilot study.

The aim of the investigators' study is to evaluate the effectiveness of nigella sativa seed in the treatment of dyslipidemia.

Dyslipidemia is a common risk factor for cardiovascular disease, the leading cause for morbidity and mortality among patients.

Nigella sativa is an easily available and acceptable remedy to treat dyslipidemia and at a low cost.

It is expected that by scientifically determining the effectiveness of this intervention it will lead to its widespread use.

This will provide a low cost alternative to treat dyslipidemia.

DETAILED DESCRIPTION:
* Pakistan is a developing country with limited resources and a high prevalence of dyslipidemia.
* Nigella sativa is a small plant originating in the Middle East and is found abundantly, growing wild in Egypt, Asiatic Turkey and the Balkan States.
* The seed extracts from this plant are used by herbalists in the treatment of several medical disorders including dyslipidemia.

OBJECTIVE:

To determine the effectiveness of the nigella sativa seed in the control of dyslipidemia in adults. This is a pilot study.

METHODOLOGY

DESIGN

Double blind, randomized, controlled trial

Inclusion Criteria:

* Adult (18 years or older) men and women who have serum cholesterol > 180 mgs/ dls
* Who consent to participate

Exclusion Criteria:

* Patients with known Diabetes Mellitus

Primary Endpoint

The primary end point for the trial is serum LDL cholesterol concentration measured at six weeks after intervention.

Secondary Endpoint

* Serum total cholesterol concentrations measured at six weeks after intervention
* Serum concentrations of HDL cholesterol measured at six weeks after intervention
* Serum concentrations of Triglyceride measured at six weeks after intervention
* Serum concentrations of Blood sugar measured at six weeks after intervention
* Changes in Serum Transminase and Serum Creatinine with six weeks of intervention

Intervention Group Recommended

* Dietary changes
* Lifestyle changes
* Nigella sativa seed as intervention.

Intervention details:

* Quantity: Two capsules of crushed nigella sativa seeds 500 mgs each
* Frequency: Twice daily
* Timing: After meals
* Duration: Six weeks

Control Group Recommended

* Dietary changes
* Lifestyle changes
* Capsules containing Calcium Lactate

Dietary Advice

Study subjects will receive advice from the Principal Investigator (PI)

* Eat low fat, low cholesterol foods
* Cut down on high fat food (fatty meats and bakery goods)
* Use low fat cooking methods (Use nonstick pans, barbecue, roast, boil)
* Avoid alcohol consumption
* Eat more fruits, vegetables and whole grains
* Subjects of both groups will be given standard low cholesterol diet sheet as well

Exercise

Subjects in both groups will be advised to take a brisk 30 minute walk for 5 days in a week on empty stomach or one hour after having a meal.

LABORATORY INVESTIGATIONS

For lab investigations venous blood specimens will be collected for the following tests. The tests will be performed on 12 hour fasting samples to assess the primary and secondary outcomes.

* Total Cholesterol
* Low Density Lipoprotein (LDL)
* High Density Lipoprotein (HDL)

Other investigations

* Triglycerides
* Fasting blood glucose (FBS)
* Creatinine SGPT (ALT)

IDENTIFICATION OF STUDY SUBJECTS

Study subjects will be identified from executive and family medicine clinics within AKUH. Individuals fulfilling the inclusion criteria will be informed about the study and asked to participate.

INFORMED CONSENT

* The participants will be informed of all possible expected benefits and possible harm ensuing from the study
* Written informed consent will be obtained from the study subjects addressing the ethical concerns of the relevant authority

RANDOMIZATION

* A randomized controlled design will be used for this trial
* Randomization will be done to give an equal chance to eligible subjects of being assigned to either group.
* A randomization plan with a block size of four will be used to assign subjects to the intervention and control groups
* This will be done in order to achieve an equal number of participants in both the groups
* A Co-Investigator will create subject identification numbers and assign group according to randomization.

FOLLOW-UP & DATA COLLECTION

* Baseline data including information on height, weight, blood pressure, blood sugar fasting, serum cholesterol, HDL, LDL, triglycerides and serum creatinine will be collected prior to starting intervention
* Subjects in both study groups will be telephoned, at an interval of 10 days by the study assistant to ensure patient compliance
* At the end of six weeks period, a fasting blood sample will be taken from the study subjects for measuring total cholesterol, LDL and HDL concentrations, serum triglycerides, blood sugar fasting and serum creatinine.
* A food diary combining groups of foods with similar nutrient content and dietary use will be given to study subjects
* Participants will record daily food intake initially and at the end of the trial period
* Patients' Body Mass Index (BMI), waist hip ratio and blood pressure will be recorded at baseline and at the end of the study.

ETHICAL ISSUES:

* Subjects in both groups of the study will be given standard dietary advice, which is recommended by National Cholesterol Education Program (NCEP) in cases fitting the inclusion criteria of this proposed study.
* In studies conducted previously, the nigella sativa seed has shown to demonstrate protective effects against nephrotoxicity and hepatotoxicity induced by either disease or chemicals.
* However, in case adverse events are observed, the intervention with nigella sativa will be stopped for that particular individual.

SAMPLE SIZE CONSIDERATIONS

This is a pilot study and will include 80 patients. Half will get N. Sativa seed capsules and the rest will get calcium lactate placebo capsules.

Analysis

* In descriptive statistics, comparison of the two treatment groups would be done on variables such as age and gender. The results will be mentioned in frequency and percentages.
* In univariate analysis t-test will be applied to detect a significant difference in the primary outcome between the two groups.
* For multivariate analysis, linear regression analysis will be used to identify variables associated with the primary outcome (LDL concentration), and to control for confounding factors. A similar process will be adopted for secondary outcome variables i.e., serum total cholesterol concentrations and HDL.

SITE

Aga Khan University Hospital (AKUH), Karachi

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years or older) men and women
* Serum cholesterol > 180 mgs/dl
* Provide Informed Consent

Exclusion Criteria:

* Diabetes mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-02; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The primary end point for the trial is serum low-density lipoprotein (LDL) cholesterol concentration measured at six weeks after intervention. | six weeks

SECONDARY OUTCOMES:
Serum total cholesterol concentrations measured at six weeks after intervention | six weeks
Serum concentrations of high-density lipoprotein (HDL) cholesterol measured at six weeks after intervention | six weeks
Serum triglyceride concentrations measured at six weeks after intervention | six weeks
Serum blood sugar concentrations measured at six weeks after intervention | six weeks
Blood pressure measured at six weeks after intervention | six weeks
Changes in serum creatinine after six weeks intervention | six weeks

CONTACTS AND LOCATIONS:
Overall Officials: Waris - Qidwai, Principal Investigator — Aga Khan University, Karachi
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Ismail J, Jafar TH, Jafary FH, White F, Faruqui AM, Chaturvedi N. Risk factors for non-fatal myocardial infarction in young South Asian adults. Heart. 2004 Mar;90(3):259-63. doi: 10.1136/hrt.2003.013631. PMID 14966040
- [Background] Ali BH, Blunden G. Pharmacological and toxicological properties of Nigella sativa. Phytother Res. 2003 Apr;17(4):299-305. doi: 10.1002/ptr.1309. PMID 12722128
- [Background] Zaoui A, Cherrah Y, Alaoui K, Mahassine N, Amarouch H, Hassar M. Effects of Nigella sativa fixed oil on blood homeostasis in rat. J Ethnopharmacol. 2002 Jan;79(1):23-6. doi: 10.1016/s0378-8741(01)00342-7. PMID 11744291
- [Background] El-Saleh SC, Al-Sagair OA, Al-Khalaf MI. Thymoquinone and Nigella sativa oil protection against methionine-induced hyperhomocysteinemia in rats. Int J Cardiol. 2004 Jan;93(1):19-23. doi: 10.1016/s0167-5273(03)00108-6. PMID 14729430
- [Derived] Qidwai W, Hamza HB, Qureshi R, Gilani A. Effectiveness, safety, and tolerability of powdered Nigella sativa (kalonji) seed in capsules on serum lipid levels, blood sugar, blood pressure, and body weight in adults: results of a randomized, double-blind controlled trial. J Altern Complement Med. 2009 Jun;15(6):639-44. doi: 10.1089/acm.2008.0367. PMID 19500003